CLINICAL TRIAL: NCT02480946
Title: A Four-Part Phase-1 Study Investigating the Tolerability, Safety and Pharmacokinetics (PK) of MBS2320 in Healthy Subjects and in Subjects With Rheumatoid Arthritis (RA) Also Treated With Methotrexate
Brief Title: Safety and Tolerability Study of MBS2320 in Healthy Subjects and Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Modern Biosciences Ltd (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 120011A; 2015-001474-18 (EudraCT Number)
Record Dates: First submitted 2015-06-16; First posted 2015-06-25 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; Osteoclastogenesis inhibitor; Anti-Inflammatory Agent; Musculoskeletal Diseases; Joint Diseases
MeSH Terms: conditions — Arthritis, Rheumatoid; Musculoskeletal Diseases; Joint Diseases | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Single Ascending Dose and Food Effect (Experimental): Part A will be a single-dose, sequential-group, double-blind, placebo-controlled study of MBS2320.
  Interventions: Drug: MBS2320; Drug: Placebo
- Multiple Ascending Dose (Experimental): Part B will be a multiple-dose, sequential-group, double-blind, placebo-controlled study to investigate 3 planned dose levels.
  Interventions: Drug: MBS2320; Drug: Placebo
- Relative Bioavailability (Experimental): Part C will be an open-label, randomised, 2-period crossover relative bioavailability study of MBS2320 in capsules or suspension. The intention is to enrol 8 healthy subjects. Each subject will participate in 2 treatment periods.
  Interventions: Drug: MBS2320; Drug: Placebo
- Drug-Drug Interaction with Methotrexate (Experimental): Part D will be a multiple dose study incorporating an open-label, fixed-sequence drug-drug interaction between MBS2320 and methotrexate and biomarker evaluation.
  Interventions: Drug: MBS2320; Drug: Methotrexate

INTERVENTIONS:
Drug: MBS2320 — As described in the arm descriptions
Drug: Placebo — As described in the arm descriptions
  Arms: Multiple Ascending Dose; Relative Bioavailability; Single Ascending Dose and Food Effect
Drug: Methotrexate — Background therapy as described in the arm descriptions
  Other Names: Rheumatrex; Trexall; Amethoperin; Mexate
  Arms: Drug-Drug Interaction with Methotrexate

SUMMARY:
Rheumatoid arthritis (RA) affects 1 percent of the population worldwide and up to 40 percent of patients don't respond to current treatments. MBS2320, the drug being tested in this trial, represents a new approach to treating RA, with the potential not only to reduce levels of inflammation but to also directly inhibit bone damage.The aim of this study is to test the safety of MBS2320 in healthy volunteers, to find out how MBS2320 levels change in the blood with dose, and to test the safety and compatibility of giving MBS2320 to patients with RA in combination with an existing treatment, methotrexate.

DETAILED DESCRIPTION:
The study will be conducted in 4 parts (parts A to D). The principal aim of this study is to obtain safety and tolerability data when MBS2320 is administered orally as single and multiple doses to healthy subjects (parts A to C). The effect of MBS2320 on the pharmacokinetics (PK) of the first-line rheumatoid arthritis (RA) therapy, methotrexate (MTX), and the effect of MTX on the PK of MBS2320, will also be evaluated in a cohort consisting of subjects with RA (Part D).

ELIGIBILITY:
Principal Inclusion Criteria:

Parts A, B, and C.

* Healthy males or females between 18 and 60 years of age.
* A body mass index (BMI) between 18.0 and 30.0 kg/m2.
* Female subjects will be of non-childbearing potential or postmenopausal as defined by the protocol.
* Female subjects must not be pregnant.

Part D

* Subjects will be otherwise healthy males or females with a diagnosis of RA between 18 and 70 years of age.
* Subjects will have a BMI between 18.0 and 30.0 kg/m2.
* Female subjects must not be pregnant.
* Subjects must have been treated with, and tolerated, oral or subcutaneous MTX for a minimum of 3 months prior to screening entry.

Principal Exclusion Criteria:

Parts A, B, and C.

* Male subjects who do not agree to use appropriate contraception.
* Female subjects who are receiving HRT who do not agree to use appropriate contraception.
* Subjects who have donated blood in the 3 months, plasma in the 7 days or platelets in the 6 weeks prior to screening.
* Subjects who consume more than the permitted alcohol requirement, who have a significant history of alcoholism or drug/chemical abuse.
* Subjects who are unwilling to abstain from alcohol as required.
* A positive urine drug screen, alcohol breath test at screening or first admission.
* Subject has received a live virus vaccination within the 30 days prior to first dose administration.
* Subjects with a positive test for tuberculosis.

Additional Part D Exclusions

* Subjects who have received any medication (except MTX) known to chronically alter drug absorption or elimination processes within 30 days prior to the first dose administration.
* Subjects currently taking any medications other than those allowed per protocol guidelines.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-07; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (incidence of all grade adverse events and dose limiting toxicities during the observation period and/or study treatment periods) | Within 7 days

SECONDARY OUTCOMES:
Study Parts A, B and C - Peak Plasma Concentration (Cmax) of MBS2320 | Part A and C - Up to 72hrs post dose, Part B - Up to 72 hrs post day 14 dose
Study Parts A, B and C - Area under the plasma concentration versus time curve (AUC) of MBS2320 | Part A and C - Up to 72hrs post dose, Part B - Up to 72 hrs post day 14 dose
Study Parts A, B and C Time to peak plasma concentration (Tmax) of MBS2320 | Part A and C - Up to 72hrs post dose, Part B - Up to 72 hrs post day 14 dose
Part D - Peak Plasma Concentration (Cmax) of MBS2320 and methotrexate | During the study treatment period
  Half-life (T1/2)
Part D - Area under the plasma concentration versus time curve (AUC) of MBS2320 and methotrexate | During the study treatment period
  Peak Plasma Concentration (Cmax), Area under the plasma concentration versus time curve (AUC), Time to peak plasma concentration (Tmax), Half-life (T1/2)
Part D - Time to peak plasma concentration (Tmax) of MBS2320 and methotrexate | During the study treatment period
Part D - Half-life (T1/2) of MBS2320 and methotrexate | During the study treatment period
Part D - Early response biomarkers of disease activity and bone turnover | Day 1 and 16.
  CRP and CTX

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, MBChB,PhD, Principal Investigator — Covance
Locations (3):
- United Kingdom (3):
  - Covance Royal Liverpool Clinical Research Unit,Royal Liverpool University Hospital, Liverpool, Merseyside
  - Covance Clinical Research Unit Ltd., Leeds, West Yorkshire
  - NIHR/Wellcome Trust Imperial Clinical Research Facility (CRF), London

IPD SHARING:
Plan to Share IPD: No